CLINICAL TRIAL: NCT06992557
Title: Clinical Evaluation of Biological Drilling Osteotomy Protocol Versus Conventional Drilling Osteotomy Protocol in the Mandibular Posterior Area a Randomized Controlled Trial
Brief Title: Clinical Evaluation of Biological Drilling Osteotomy Protocol Versus Conventional Drilling Osteotomy Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mazen Mostafa Sayed, Assistant lecturer in The General Organization for Teaching Hospitals and Institutes, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mazenmostafasayedali@@15121987
Record Dates: First submitted 2025-05-12; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Implant Stability; Low Speed Drilling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biological drilling osteotomy protocol (Experimental): * Local infiltration anesthesia will be applied to all the patients participating in this study.
  * Full thickness mucoperiosteal flap reflection with 15c blade.
  * Osteotomy site preparation through sequential biologic drilling in healed bony site with a pilot drill at 800 rpm with irrigation initiates the drilling process, which is then followed by drills of different sizes and shapes at low speeds at 150rpm without irrigation.
  * The implant will be positioned in the osteotomy site and a healing collar will be placed.
  * The mucoperiosteal flap will be sutured in an interrupted manner with 5-0 proline suture material
  Interventions: Procedure: Biological drilling osteotomy protocol
- Conventional drilling osteotomy protocol (Active Comparator): * Local infiltration anesthesia will be applied to all the patients participating in this study.
  * Full thickness mucoperiosteal flap reflection with 15c blade.
  * Preparation for osteotomy site with conventional sequential drilling in healed bony site at 1200 rpm with irrigation.
  * The implant will be positioned in the osteotomy site and a healing collar will be placed.
  * The mucoperiosteal flap will be sutured in an interrupted manner with 5-0 proline suture material.
  Interventions: Procedure: Conventional drilling osteotomy protocol

INTERVENTIONS:
Procedure: Biological drilling osteotomy protocol — * Osteotomy site preparation through sequential biologic drilling in healed bony site with a pilot drill at 800 rpm with irrigation initiates the drilling process, which is then followed by drills of different sizes and shapes at low speeds at 150rpm without irrigation.
  * The implant will be positioned in the osteotomy site and a healing collar will be placed.
  Arms: Biological drilling osteotomy protocol
Procedure: Conventional drilling osteotomy protocol — * Preparation for osteotomy site with conventional sequential drilling in healed bony site at 1200 rpm with irrigation.
  * The implant will be positioned in the osteotomy site and a healing collar will be placed.
  Arms: Conventional drilling osteotomy protocol

SUMMARY:
This study aims to evaluate the effect of biological drilling osteotomy protocol compared to conventional osteotomy protocol in delayed implant placement in the posterior mandible regarding implant stability Type of study design: Randomized Clinical Trial In patient indicated for delayed implant placement in the lower posterior mandible will the use of biological drilling protocol osteotomy compared to conventional drilling protocol osteotomy differ regarding implant stability at three months?

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy male and female patients, aged 21 to 60 years old,
* Indicated for delayed implant placement in the posterior mandibular arch.
* Good oral health.
* Willingness to sign the informed consent form.

Exclusion Criteria:

* Heavy smoker (> 10 cigarettes/day)
* Pregnant females
* Contraindication for Implant surgery.
* Patients with poor oral hygiene.
* A history of radiotherapy in the head or neck region.
* Patients with systemic disease like uncontrolled diabetes mellitus, coagulation disorders, alcohol or drug abuse not suitable for implantation.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Implant stability (Implant Stability Quotient ) | Measurements will be taken immediately post surgical ,3 weeks,2 month and 3 months post surgical
  Scale ranges from 1 to 100, the higher the Implant stability quotient the more stability

SECONDARY OUTCOMES:
Crestal bone level changes | Measurements will be taken immediately post surgical and after 3 months post surgical
  Long-cone intraoral radiographs were collected under controlled circumstances with personalised X-ray holders (XPC) and a registration bite block for repeatable imaging. The periapical radiographs carried out by digital sensor size 2 standardized film and standardized exposure settings The neck of the implant was taken as a reference point in all images for standardization post surgically and after 3 months.
Post-Operative Pain ( visual analogue scale) | 7 days post surgically
  Filled in by the patient after being given instructions about charting by the dental operator
Post-operative swelling (Verbal rating scale) | Swelling will be assessed 7 days post surgically
  Filled in by the patient after being given instructions about charting by the dental operator.
  * Absent(no swelling)
  * Slight (intraoral swelling at the operated area)
  * Moderate (moderate intraoral swelling at the operated area)
  * Intense (intensive extra oral swelling extending beyond the operated area).
Post-Operative patient's Satisfaction | 3 months post surgically
  Three Yes or No Questions will be asked to the patient about his overall satisfaction about the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university , faculty of dentistry, Cairo, Egypt